CLINICAL TRIAL: NCT06430320
Title: Long Term Effectiveness of Uterine Sparing Fibroid Treatments
Brief Title: Ascertaining Longterm Outcomes of Fibroid Treatments
Acronym: ALOFT
Status: Enrolling by invitation | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Mayo Clinic (Other); University of California, San Francisco (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Lisa King, Principal Investigator, Henry Ford Health System
Other Study IDs: R9NXPE2GTCN9
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Uterine Fibroid
Keywords: Uterine fibroid treatment; Multi-center, prospective, observational cohort study; Uterine-sparing treatment procedures; Patient-reported outcomes; Quality of life
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: NA- no intervention — NA- no intervention

SUMMARY:
The goal of the ALOFT study is to understand the health of women in the 12 years following a uterine fibroid (UF) treatment. ALOFT is a multi-center, prospective, observational cohort study of approximately 700 women who have undergone uterine-sparing treatment procedures for UF and previously participated in the longitudinal studies COMPARE-UF (NCT02260752) or ULTRA (NCT02100904).

The primary uterine sparing treatment procedures undergone by study participants are myomectomy, endometrial ablation (EA), uterine artery embolization (UAE) and laparoscopic radiofrequency ablation (RFA). A smaller number of women may be studied who underwent focused ultrasound, intrauterine device (IUD), and medical management.

Two follow-up study contacts with COMPARE-UF and ULTRA participants will occur to assess changes in UF symptoms and treatment failure which is defined as the need for another UF treatment procedure. Questionnaires will be used to collect data on patient-reported characteristics and outcomes and quality of life.

The study's analyses will focus on comparisons of primary and secondary outcomes among women.

ELIGIBILITY:
Inclusion Criteria:

* Participant has to have been enrolled in either the COMPARE-UF or ULTRA study
* Participant had a uterine-sparing fibroid treatment at enrollment in COMPARE-UF or ULTRA study

Exclusion Criteria:

* Individuals who were not consented into the original COMPARE-UF or ULTRA study
* Individuals who did not have a uterine-sparing fibroid treatment at enrollment in COMPARE-UF or ULTRA study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Participants who were previously enrolled in either the COMPARE-UF or ULTRA study
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure | Up to 12 years
  The need for another uterine fibroid treatment procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ganesa Wegienka, PhD, Principal Investigator — Henry Ford Health
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Henry Ford Health, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ALOFT study landing page — https://www.henryford.com/hcp/research/aloft-study